CLINICAL TRIAL: NCT02094599
Title: A Single-dose, Double-blind, Double-dummy, Randomized, Placebo- and Active-controlled Crossover Study to Evaluate the Abuse Potential of Dronabinol Oral Solution in Recreational Cannabinoid Users
Brief Title: A Study of the Abuse Potential of Dronabinol in Recreational Cannabinoid Users
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: INSYS Therapeutics Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Triple
Other Study IDs: INS-13-017
Record Dates: First submitted 2014-03-14; First posted 2014-03-24 (Estimated); Last update posted 2014-05-13 (Estimated); Status verified 2014-05

CONDITIONS: Drug Abuse, Medication
MeSH Terms: conditions — Substance-Related Disorders | interventions — Dronabinol

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor

ARMS (1):
- All Enrolled Participants (Experimental): Each participant receives all treatments (of placebo, dronabinol 10 mg and dronabinol 30 mg) in a 5-way crossover design. At each treatment visit, participants receive a single dose, contained in two syringes of oral solution and three capsules. When dronabinol is in syringes, placebo is in capsules, and when dronabinol is in capsules, placebo is in syringes. When assigned to take placebo only, placebo is in both the syringes and the capsules.
  Interventions: Drug: Dronabinol 10 mg; Drug: Dronabinol 30 mg; Drug: Placebo

INTERVENTIONS:
Drug: Dronabinol 10 mg — Dronabinol at a strength equivalent to 10 mg provided in capsules or as an oral solution in syringes.
Drug: Dronabinol 30 mg — Dronabinol at a strength equivalent to 30 mg provided in capsules or as an oral solution in syringes.
Drug: Placebo — Matching placebo provided in capsules or as an oral solution in syringes.

SUMMARY:
The primary objective of this study is to evaluate the abuse potential of dronabinol oral solution in recreational cannabinoid users.

DETAILED DESCRIPTION:
Following a four-day period for screening and qualification, there are five treatment visits with a minimum 8-day washout between treatments. Each participant will receive all treatments in a 5-way crossover design.

ELIGIBILITY:
Inclusion Criteria:

* Healthy adult protocol-defined recreational cannabinoid user
* Meets protocol-specified criteria for qualification and contraception
* Able to speak, read and understand English well enough to understand the nature of the study, provide written informed consent, and to allow completion of all study assessments
* Provides written informed consent prior to any protocol-specific procedures, and agrees to abide by all protocol-specified requirements and restrictions

Exclusion Criteria:

* Dependence on any substance other than nicotine or caffeine beyond protocol-specified limits
* Signs, symptoms or history of any condition that, per protocol or in the opinion of the investigator, might compromise: 1) the safety or well-being of the participant or study staff, 2) the safety or well-being of the participant's offspring (such as through pregnancy or breast-feeding), 3) the analysis of results
* Unwilling, unable, or unlikely to follow protocol-specified restrictions on food, drink, nicotine or physical activities (such as exercise and driving)
* An employee of the sponsor or research site personnel directly affiliated with this study or their immediate biological or adopted family member defined as a spouse, parent, child or sibling

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 43 (Actual)
Dates: Start 2014-02; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
Peak score (Emax) on Drug Liking calculated from a 100-point visual analogue scale (VAS), where 0=strong disliking and 100=strong liking | within 24 hours post-dose

SECONDARY OUTCOMES:
Peak score (Emax) for Drug Effects, calculated from scores on a VAS scale of 0-100, where 0=not at all and 100=extremely | within 24 hours post-dose
  Categorical measures = Good drug effects, High, Stoned, Bad effects, Any effects
Peak score (Emax) for a shortened Addiction Research Center Inventory (ARCI) scale of 0-49, where 49 is the highest possible score | within 24 hours post-dose
  Categorical measures = Euphoria, Dysphoria, Sedation, Marijuana
Peak score (Emax) for Subjective Drug Value (SDV) in dollars | within 24 hours post-dose
Time-averaged Area under the Effect Curve (TA_AUC) for Drug Effects, calculated from scores on a VAS scale of 0-100, where 0=not at all and 100=extremely | within 24 hours post-dose
  Categorical measures = Good drug effects, High, Stoned, Bad effects, Any effects
Overall Drug Liking (Emax/Emin) calculated from a 100-point visual analogue scale (VAS), where 0=strong disliking and 100=strong liking | within 24 hours post-dose
Time-averaged Area under the Effect Curve (TA_AUC) for Drug Liking calculated from a 100-point visual analogue scale (VAS), where 0=strong disliking and 100=strong liking | within 24 hours post-dose
Time-averaged Area under the Effect Curve (TA_AUC) for a shortened Addiction Research Center Inventory (ARCI) scale of 0-49, where 49 is the highest possible score | within 24 hours post-dose
  Categorical measures = Euphoria, Dysphoria, Sedation, Marijuana
Trough Score (Emin) for Drug Liking calculated from a 100-point visual analogue scale (VAS), where 0=strong disliking and 100=strong liking | within 24 hours post-dose
Peak score (Emax) for Take Drug Again, calculated from scores on a VAS scale of 0-100, where 0=definitely not and 100=definitely so | within 24 hours post-dose
Peak score (Emax) for Alertness/Drowsiness, calculated from scores on a VAS scale of 0-100, where 0=very drowsy and 100=very alert | within 24 hours post-dose
Time-averaged Area under the Effect Curve (TA_AUC) for Alertness/Drowsiness, calculated from a 100-point visual analogue scale (VAS), where 0=very drowsy and 100=very alert | within 24 hours post-dose

CONTACTS AND LOCATIONS:
Overall Officials: Larry Dillaha, MD, Study Director — INSYS Therapeutics Inc; Michael McDonnell, MD, Principal Investigator — INC Research Toronto, Inc.
Locations (1):
- INC Research Toronto, Inc., Toronto, Ontario, Canada